CLINICAL TRIAL: NCT04585464
Title: A Phase 1, Randomized, Placebo-Controlled, Double-blind, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and PK of EDG-5506 in Adult Healthy Volunteers and Adults With Becker Muscular Dystrophy
Brief Title: A Study to Assess Safety, Tolerability, and PK of EDG-5506 in Healthy Volunteers and Becker Muscular Dystrophy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Edgewise Therapeutics, Inc. (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EDG-5506-001
Record Dates: First submitted 2020-10-02; First posted 2020-10-14 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Healthy Volunteer; Becker Muscular Dystrophy
Keywords: Healthy Volunteers; Becker Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Healthy Volunteer: Single Ascending Dose (Experimental): Single oral ascending dose in healthy volunteers
  Interventions:
  Drug: EDG-5506 Drug: Placebo
  Interventions: Drug: EDG-5506; Drug: Placebo
- Healthy Volunteer: Multiple Ascending Dose (Experimental): Multiple oral ascending doses in healthy volunteers
  Interventions:
  Drug: EDG-5506 Drug: Placebo
  Interventions: Drug: EDG-5506; Drug: Placebo
- Becker Muscular Dystrophy: Multiple Ascending Dose (Experimental): Multiple oral ascending doses in adults with Becker muscular dystrophy
  Interventions:
  Drug: EDG-5506 Drug: Placebo
  Interventions: Drug: EDG-5506; Drug: Placebo

INTERVENTIONS:
Drug: EDG-5506 — EDG-5506 is administered orally as a single dose or once daily
Drug: Placebo — Placebo is administered orally as a single dose or once daily

SUMMARY:
EDG-5506 is an investigational product intended to protect and improve function of dystrophic muscle fibers. This Phase 1 study of EDG-5506 will assess the safety, tolerability, and pharmacokinetics (PK) and of EDG-5506 in adult healthy volunteers and in adults with Becker muscular dystrophy (BMD).

DETAILED DESCRIPTION:
Enrolled participants in this study will receive a single oral dose or multiple oral doses of EDG-5506 or a placebo. Blood and urine samples will be collected to measure how EDG-5506 is processed by the body and how the body responds when exposed to EDG-5506. Participants in the single ascending dose part of the study will remain in the clinic for 7 days with a 42-day follow-up period. Participants in the multiple ascending dose part of the study will remain in the clinic for 16 days with a 13-day follow-up period. Safety, tolerability, and pharmacokinetics of EDG-5506 will be assessed in healthy volunteers prior to enrolling participants with Becker muscular dystrophy.

ELIGIBILITY:
Inclusion Criteria:

* For all potential participants (Healthy volunteers and BMD): Male or for HV: female. For all: adults aged 18 to 55 years at time of consent.
* For HVs: Good general health, with no significant medical history, no clinically significant abnormalities on physical exam
* For BMD: Diagnosis of BMD based on documentation of mutation(s) in the dystrophin gene and BMD phenotype
* For BMD: Ability to ambulate
* For all: Weight greater than or equal to 50 kg and BMI less than 33 kg/m2
* For HV: Females must be of non-childbearing potential.
* For all: Males with female partners must use a medically accepted contraceptive regimen from first dose through 90 days after the last dose
* For all: Non-smoker and must not have used any tobacco products within 3 months prior to the Screening visit.
* For all: Able and willing to attend the necessary visits at the study center.

Exclusion Criteria:

* For all: History of, or physical exam findings indicating clinically significant endocrine, neurological, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases that, in the opinion of the Investigator, would render the subject being unsuitable for the study.
* For all: Unable to refrain from strenuous exercise for 3 days prior to check-in and during study.
* For all: Participation in any other investigational drug study within 30 days or 5 half-lives (whichever is longer) of dosing in the present study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy volunteers: Male and non-childbearing potential females. Male Becker muscular dystrophy (BMD) participants
Enrollment: 127 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-12-27 (Actual)

PRIMARY OUTCOMES:
Incidence, frequency, severity and dose-relationship of adverse events | Up to 42 days of monitoring
Incidence of abnormal laboratory test results (clinical chemistry, hematology, urinalysis, coagulation) | Up to 42 days of monitoring
Incidence of treatment-emergent clinically abnormal electrocardiogram (ECG) | Up to 42 days of monitoring
Incidence of abnormal vital signs | Up to 42 days of monitoring
Incidence of abnormal physical exam findings | Up to 42 days of monitoring

SECONDARY OUTCOMES:
Plasma maximum measured drug concentration (Cmax) | Up to 42 days of testing
Time of maximum concentration (Tmax) | Up to 42 days of testing
Area under the concentration-time curve (AUC) | Up to 42 days of testing
Plasma half-life (T½) | Up to 42 days of testing
Renal clearance (CLR) | Up to 42 days of testing
Drug excreted unchanged in urine (Amt0-24) | Up to 42 days of testing
Fraction excreted in urine (Fe) | Up to 42 days of testing

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Edgewise Therapeutics, Inc.
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Donovan J, Silverman JA, Barthel B, DuVall M, Madden M, MacDougall J, Kilburn NR, Bronson A, Evanchik M, Gordon G, Koch K, Russell AJ. A Phase 1, Double-Blind, Placebo-Controlled Trial of Sevasemten (EDG-5506), a Selective Modulator of Fast Skeletal Muscle Contraction, in Healthy Volunteers and Adults With Becker Muscular Dystrophy. Muscle Nerve. 2025 Sep;72(3):399-407. doi: 10.1002/mus.28444. Epub 2025 Jun 2. PMID 40452637
- See also: Sponsor Website — http://www.edgewisetx.com